CLINICAL TRIAL: NCT05176756
Title: A Randomized Controlled Trial of Strategies to Augment Physical Activity in Black and Hispanic Breast and Prostate Cancer Survivors (ALLSTAR)
Brief Title: RCT of Strategies to Augment Physical Activity in Black and Hispanic Breast and Prostate Cancer Survivors (ALLSTAR)
Acronym: ALLSTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: American Heart Association (Other); City of Hope National Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UPCC 21921; 849679 (Other: University of Pennsylvania)
Record Dates: First submitted 2021-12-15; First posted 2022-01-04 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases; Breast Cancer; Prostate Cancer; Physical Inactivity
Keywords: physical activity; cardiovascular disease; randomized controlled trial; breast cancer; prostate cancer
MeSH Terms: conditions — Cardiovascular Diseases; Breast Neoplasms; Prostatic Neoplasms; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Attention Control (Active Comparator): In addition to using a wearable device, participants in this arm will receive a daily notification of their step count from the previous day. This notification serves as an 'attention control' and allows us to better isolate the impact of the gamification with social support. It may also help to reduce differential attrition across arms.
  Interventions: Behavioral: Attention control
- Gamification and Social Support (Experimental): Participants in this arm will receive the same devices and daily messaging as control. They will also be entered into a game designed using behavioral economic principles for 6 months. This intervention has been adapted from our prior successful pilot studies. The game runs automatically and does not require any effort on the part of the participant to 'play' the game other than to strive for physical activity goals. Participants in this arm will also select a family member or friend who will serve as a support partner to encourage the participant to meet their step goals. The gamification and social support interventions will end after 6 months at which point participants will receive the same treatment as the attention control arm for the 3-month follow-up period.
  Interventions: Behavioral: Gamification and Social Support

INTERVENTIONS:
Behavioral: Gamification and Social Support — Participants will be entered into a points and levels-based game designed to help them meet their step count goals. At the start of each week, the participant will receive a set amount of points. Each day their step goal is not met, they lose points. If the participant meets a certain point value at the end of the week, they will either advance one level (of five total levels); if they do not, they will drop one level. Each participant will also select a family member or friend or the study coordinator to serve as a support partner. At the beginning of the intervention, the participant and support partner will identify at least 3 ways in which they can help the participant meet their step goals. This partner will receive a weekly email reminding them of these approaches and updating them on the participant's progress.
  Arms: Gamification and Social Support
Behavioral: Attention control — Participants will receive a daily text message with their step count from the day prior.
  Arms: Attention Control

SUMMARY:
This is a two-arm, randomized, controlled trial to evaluate the effectiveness of using a behaviorally designed gamification intervention with social support compared to an attention control group to increase physical activity during a 6-month intervention with a 3-month follow-up period. We will enroll 150 Black or Hispanic breast and prostate cancer survivors who are at an especially high risk for developing major CVD from two U.S. cancer centers: the University of Pennsylvania Health System and City of Hope National Medical Center. All participants will receive a wearable activity tracker (Fitbit) and will be enrolled in the Way to Health system, a research information technology platform at the University of Pennsylvania. Within the Way to Health platform, patients will set a goal to increase daily step count from baseline, and will then be randomized to gamification plus social support or to attention control. The study will evaluate the effect of the gamification intervention on daily physical activity (as measured by daily steps and moderate to vigorous physical activity), physical function, fatigue, and health-related quality of life.

DETAILED DESCRIPTION:
The specific objectives of this study are the following:

1. To determine the effectiveness of a behaviorally designed gamification intervention with social support to increase physical activity in Black and Hispanic breast and prostate cancer survivors
2. To evaluate the effects of the gamification intervention on physical function, fatigue, and health-related quality of life

Recruitment: Participants will be recruited from the tumor registries at the two cancer centers or via direct referral from these two health systems. Patients identified from tumor registries will be emailed a link to the study, after obtaining provider permission to contact. Patients will then be contacted by phone two weeks later to further discuss the study. Interested patients will visit the study website on the Way to Health platform to learn more about the study, create an account, provide informed consent, and complete initial baseline eligibility surveys. Study coordinators will be available to assist patients with this process, as necessary.

Informed Consent: We will follow an IRB-approved approach taken by many studies using the Way to Health platform to obtaining informed consent. Upon reaching the portal, potential participants will be asked to create an account and will then be informed of the details of the study, including its objectives, duration, requirements, and financial payments. The Way to Health portal will then take interested participants through an online informed consent. Successive screens will explain the voluntary nature of the study, the risks and benefits of participation, alternatives to participation, and that participants can withdraw from the study at any time. On the final consent screen, potential participants who click a clearly delineated button stating that they agree to participate in the study will be considered to have consented to enroll. Participants will be provided with details regarding how to contact the research team via email or phone at any time if they subsequently wish to withdraw from the study. Support partners will provide verbal informed consent via telephone for their name, email address, and phone number to be stored in the study database. For participants who are English-speaking but illiterate, an authorized family member will be present to witness the oral presentation of the consent form and both participant and authorized family member sign the consent form. Spanish speaking patients will be consented with the aid of a medical interpreter. Directly referred patients will also complete informed consent via the Way to Health platform as above.

Enrollment: Immediately after completing the informed consent process, potentially eligible patients will be prescreened to ensure they meet the eligibility criteria. Simultaneously, participants will complete an online questionnaire to confirm eligibility and complete the study surveys.

Study surveys: The baseline questionnaire will include demographics, as well as validated surveys on health status, exercise self-efficacy, other forms of exercise besides step counts (e.g. swimming, biking), and health-related quality of life (EQ-5D-5L). To assess physical function and fatigue, they will complete the Patient Reported Outcome Measure Information System (PROMIS) Physical Function, Global-10 scales, 6b, and Cancer Fatigue Short Form scales. We will also assess the social determinants of health (SDOH) through a validated, reliable and reproducible instrument focused on the core, structural, and individual SDOH.

Determination of Baseline Step Count and Goal-Setting: After completing the baseline questionnaire, eligible participants will be mailed a wearable activity tracking device and asked to get used to the wearable device for a few weeks. During this run-in period, baseline activity measures (daily step counts, minutes of moderate-to-vigorous physical activity, minutes of sleep) will be estimated. If fewer than 4 days of data are available during the second week, study coordinators will reach out to the participant to inquire about any device issues and the run-in period will be extended until at least 4 days of data are captured. Participants who do not complete this run-in phase will not be randomized into the trial, nor will patients with step counts > 7500 steps/day during the run-in phase. Once baseline measures have been established, eligible participants will be contacted to choose a goal step goal increase between 1500 to 3000 steps above their baseline. Participants will be able to adjust their step goal at any time during the study, as long as it is within this range.

Randomization: Participants that have established baseline measures and finished goal selection will be randomly assigned to control or the intervention using a 1:1 allocation, stratifying by site (Penn or City of Hope) and on baseline step count (<4000, 4000-5999, 6000-7500), and block sizes of 2 using an electronic number generator through the Way to Health platform.

End-of-study: At the end of the 6-month intervention and 3-month follow-up period, patients will be alerted by the Way to Health platform to return to the study website to complete an end-of-study questionnaire consisting of the EQ-5D-5L, PROMIS Physical Function and Global-10 scales, the PROMIS Cancer Fatigue Short Form, and the Godin Leisure Time exercise questionnaire.

Subject compensation: To reduce dropout and the risk of differential attrition by arm, all participants will receive $25 for enrolling in the study, $25 for completing 6-months, and $50 for completing 9 months (total of $100).

Data analyses: Data for all consented patients, whether or not they completed all protocol requirements, will be included for analysis. All analyses will be performed by faculty and staff statisticians at the University of Pennsylvania using intention-to-treat and will be adjusted for the stratification factors used at randomization. A two-sided Type I error=0.05 will be used.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with breast or prostate cancer and treated with cardiotoxic therapy (e.g. anthracyclines, chest radiation, trastuzumab, aromatase inhibitors, or ADT)
* Have ≥1 cardiovascular risk factors (e.g. hypertension, diabetes, dyslipidemia, obesity) or known coronary artery disease (prior coronary revascularization, myocardial infarction, or coronary stenosis > 70%), or are 65+ years of age at time of enrollment
* Self-identify as Black or Hispanic
* Are at least 2 years from their cancer diagnosis and have no evidence of active malignancy or acute illness that would limit study participation
* Own a smartphone or tablet compatible with the wearable device
* Are able to read English or Spanish
* Are able to provide informed consent

Exclusion Criteria:

* Currently participating in another physical activity research study
* Have any medical conditions prohibiting ambulation without assistance
* Any other reason why it is not feasible or safe to complete the entire 9-month study
* Step count > 7500/day during the baseline data collection period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Change in daily step count | Baseline to the 6-month intervention period
  Change in daily step count for patients in intervention arm versus patients in the attention control arm

SECONDARY OUTCOMES:
Change in daily step count | Baseline to the 3-month follow-up period
  Change in daily step count for patients in intervention arm versus patients in the attention control arm
Change in daily minutes of moderate or vigorous physical activity (MVPA) | Baseline to the 6-month intervention period
  Change in daily minutes of moderate or vigorous physical activity in patients in intervention arm versus patients in the attention control arm
Change in daily minutes of moderate or vigorous physical activity (MVPA) | Baseline to the 3-month follow-up period
  Change in daily minutes of moderate or vigorous physical activity in patients in intervention arm versus patients in the attention control arm

OTHER OUTCOMES:
Change in PROMIS Physical Function 6b scale | Baseline to the 6-month intervention period
  Change in PROMIS Physical Function 6b scale in patients in intervention arm versus patients in the attention control arm
Change in PROMIS Physical Function 6b scale | Baseline to the 3-month follow-up period
  Change in PROMIS Physical Function 6b scale in patients in intervention arm versus patients in the attention control arm
Change in PROMIS Cancer Fatigue Short Form | Baseline to the 3-month follow-up period
  Change in PROMIS Cancer Fatigue Short Form in patients in intervention arm versus patients in the attention control arm
Change in PROMIS Cancer Fatigue Short Form | Baseline to the 6-month intervention period
  Change in PROMIS Cancer Fatigue Short Form in patients in intervention arm versus patients in the attention control arm
Change in EQ-5D-5L | Baseline to the 6-month intervention period
  Change in EQ-5D-5L in patients in intervention arm versus patients in the attention control arm
Change in EQ-5D-5L | Baseline to the 3-month follow-up period
  Change in EQ-5D-5L in patients in intervention arm versus patients in the attention control arm

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, MD, PhD, Principal Investigator — University of Pennsylvania; Alexander C. Fanaroff, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - City of Hope National Medical Center, Duarte, California
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fanaroff AC, Orr JA, Anucha C, Kim E, Rareshide C, Zhu J, Echevarria M, Rodarte S, Kassabian M, Balasian E, Ky B, Volpp KG, Armenian SH. Behaviorally Designed Gamification and Physical Activity Among Breast and Prostate Cancer Survivors. JACC CardioOncol. 2025 Nov 3:S2666-0873(25)00348-5. doi: 10.1016/j.jaccao.2025.10.001. Online ahead of print. PMID 41182202
- [Derived] Fanaroff AC, Orr JA, Anucha C, Kim E, Rareshide C, Echevarria M, Rodarte S, Kassabian M, Balasian E, Ky B, Volpp KGM, Armenian S. A randomized controlled trial of gamification to increase physical activity among black and Hispanic breast and prostate cancer survivors: Rationale and design of the ALLSTAR clinical trial. Am Heart J. 2025 Feb;280:42-51. doi: 10.1016/j.ahj.2024.10.021. Epub 2024 Nov 4. PMID 39505121
- [Derived] Barrett M, Wilcox NS, Huang A, Levy R, Demissei B, Narayan V, Ky B. Bearing allostatic load: insights into a more equitable future within cardio-oncology. Trends Mol Med. 2022 Dec;28(12):1040-1049. doi: 10.1016/j.molmed.2022.09.006. Epub 2022 Oct 4. PMID 36207229